CLINICAL TRIAL: NCT03028610
Title: Pregnancy Outcome Following Global Fibroid Ablation Using the Acessa™ System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFA-001
Record Dates: First submitted 2016-08-02; First posted 2017-01-23 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: One or More Uterine Fibroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acessa™ System (Experimental): radiofrequency generator
  Interventions: Device: radiofrequency generator

INTERVENTIONS:
Device: radiofrequency generator

SUMMARY:
Prospective, interventional, single-center, longitudinal, single-arm pilot study to evaluate pregnancies following the Acessa™ treatment of uterine myomas in women who desire future childbearing

ELIGIBILITY:
Inclusion Criteria:

1. Are premenopausal and aged 18 to 40 years.
2. Have already consented to have their fibroids treated with the Acessa™ procedure.
3. Desire pregnancy within two years following Acessa™ treatment
4. Have a normal endometrial cavity as delineated by sonohysterogram within 6 months prior to treatment.
5. Have a uterine size relating to ≤14 weeks of pregnancy, as determined by palpatory pelvic exam.
6. Have fibroids identified by transvaginal ultrasound with:

   1. ≤6 (six) fibroids of ≤5 cm at the major diameter
   2. a total uterine volume of no greater than 300 cc
7. Patients with type 2 fibroids are acceptable for inclusion.
8. Are current in their screening for cervical cancer precursors (i.e. PAP 1 or 2).
9. Are capable of providing informed consent.
10. Are willing and able to comply with all study tests, procedures, and assessment tools during screening and up to 3 years post treatment.
11. Are able to pass a pre-operative health exam (ASA I-III).
12. Patients who are currently undergoing fertility treatments (e.g. Clomid, IVF, etc.) or who are planning such treatments may be enrolled in the study.

Exclusion Criteria:

1. Have contraindications for laparoscopic surgery and/or general anesthesia.
2. Have cervical myomas or Type 0 or Type 1 myomas. Type 0 and Type 1 myomas are excluded as these are generally accessible to hysteroscopic approaches. Cervical myomas are difficult to treat and present a greater risk of bladder or urethral injury.
3. Have one or more Type 0 (completely intracavitary) or Type 1 resectable submucous fibroids.
4. Have known or suspected abdominal adhesions which are expected to complicate laparoscopic surgery.
5. Have known or suspected untreated intra-uterine adhesions or uterine septum.
6. Have previously undergone endometrial ablation, uterine artery embolization, or uterine artery ligation/occlusion, high-intensity focused ultrasound, laparoscopic, hysteroscopic or abdominal myomectomy, or any other uterine-preserving technique for reduction of menstrual bleeding.
7. Subjects taking platelet-inhibiting drugs such as nonsteroidal anti-inflammatory drugs (NSAIDs), aspirin, and clopidogrel
8. Are pregnant or lactating.
9. Have known or suspected severe endometriosis.
10. Have known or suspected adenomyosis.
11. Have active or history of pelvic inflammatory disease.
12. Have a history of or evidence of gynecologic malignancy or pre-malignancy within the past five years.
13. Have had pelvic radiation.
14. Have a persistent and undiagnosed complex adnexal mass.Are unable to give informed consent.
15. In the medical judgment of the investigator should not participate in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
Spontaneous abortion | 6 months
Ectopic pregnancy | three years
Vaginal delivery and either | three years
  i. Uncomplicated delivery or ii. Delivery with complications such as:
  * Premature rupture of the membranes (PROM) or
  * Preterm premature rupture of the membranes (PPROM)
Caesarean section delivery and either | three years
  i. Uncomplicated delivery or ii. Delivery with complications such as:
  * Preterm delivery
  * Preterm labor
  * Uterine rupture
  * Stillbirths
  * Postpartum

SECONDARY OUTCOMES:
Procedure-related complications within 1 month post-procedure | 1 month
Post-treatment readmission and reintervention rate within 1 month post-procedure assessed by questionnairie | 1 month
Post-treatment changes in menstrual status up to 36 months post-procedure assessed by a menstrual impact score | three years
Post-treatment changes in myoma size as determined by ultrasound | 3, 6, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Sara Y Brucker, MD, Principal Investigator — University Women's Hospital, Calwerstrasse 7, 72076 Tübingen, Germany
Locations (1):
- University Women's Hospital, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No